CLINICAL TRIAL: NCT06761001
Title: Investigation of the Effect of I-PRF Application on Pain in Alveolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Gorkem Tekin, Asst.Prof., Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EskisehirOU-TEKIN-001
Record Dates: First submitted 2024-12-30; First posted 2025-01-07 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Alveolar Osteitis; Pain; Dry Socket
Keywords: injectable platelet rich fibrine
MeSH Terms: conditions — Dry Socket; Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-PRF (Experimental): I-PRF Application
  Interventions: Device: I-PRF
- Standard treatment (Active Comparator): standard treatment
  Interventions: Other: Control

INTERVENTIONS:
Device: I-PRF — After local anesthesia is injected, alveolar curettage is performed and the socket is irrigated with saline solution. I-PRF is given to patients in the experimental group.
  Arms: I-PRF
Other: Control — After local anesthesia is injected, alveolar curettage is performed and the socket is irrigated with saline solution.
  Arms: Standard treatment

SUMMARY:
Literature review showed that there are no studies on the use of i-PRF in alveolitis cases. The aim of this study was to investigate the effect of i-PRF on the treatment of alveolitis. The hypothesis of the study was that i-PRF applied to alveolitis patients would reduce pain.

DETAILED DESCRIPTION:
The present study will include 60 healthy patients over 18 years of age with alveolitis. 60 patients will be randomly divided into two groups: Control and I-PRF. After irrigation of the sockets, no substance will be applied to the control group, and I-PRF will be applied to the study group. Postoperative pain will be measured on the 3rd and 7th days.

ELIGIBILITY:
Inclusion Criteria:

Healthy individuals without systemic disease Patients with complete data and attending their appointments

Exclusion Criteria:

Patients who smoke Pregnant or breastfeeding female patients with bleeding disorders and diabetics Patients currently or previously using bisphosphonates or receiving radiotherapy to the jaw Patients unable to consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-20 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Change in post-operative pain assessed: visual analog (VAS) scale | postoperative 3rd, and 7th days
  VAS measured on a 10cm scale, where 0 represents no pain and 10 represents maximum pain

CONTACTS AND LOCATIONS:
Overall Officials: Görkem TEKİN, Assist.Prof., Study Chair — Eskişehir Osmangazi University Faculty of Dentistry
Locations (1):
- Eskişehir Osmangazi University, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD may share with other researchers upon request

REFERENCES:
- [Result] Uranbey O, Ayranci F. How effective are concentrated growth factor and injectable platelets in reducing complications following impacted third molar surgery? Quintessence Int. 2024 May 30;55(5):380-390. doi: 10.3290/j.qi.b5213477. PMID 38619256
- [Result] Laforgia A, Inchingolo AD, Riccaldo L, Avantario P, Buongiorno S, Malcangi G, Bordea IR, Palermo A, Inchingolo F, Inchingolo AM, Dipalma G. The Use of Platelet-Rich Fibrin (PRF) in the Management of Dry Socket: A Systematic Review. Int J Mol Sci. 2024 Sep 19;25(18):10069. doi: 10.3390/ijms251810069. PMID 39337554
- [Result] Sharma A, Aggarwal N, Rastogi S, Choudhury R, Tripathi S. Effectiveness of platelet-rich fibrin in the management of pain and delayed wound healing associated with established alveolar osteitis (dry socket). Eur J Dent. 2017 Oct-Dec;11(4):508-513. doi: 10.4103/ejd.ejd_346_16. PMID 29279679
- [Derived] Tekin G, Turedi SO. Is injectable platelet-rich fibrin really effective in alveolar osteitis? a randomised controlled clinical trial. BMC Oral Health. 2025 May 26;25(1):804. doi: 10.1186/s12903-025-06257-y. PMID 40420265